CLINICAL TRIAL: NCT02475343
Title: A Novel Method to Assess the Cornea Biomechanical Properties With Schiotz
Brief Title: A Novel Method to Assess the Cornea Biomechanical Properties With Schiotz Tonometer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhiwei Li (Other Government)
Responsible Party: Sponsor-Investigator, Zhiwei Li, Dr., Shandong Provincial Hospital
Organization: Shandong Provincial Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: No.018
Record Dates: First submitted 2015-05-28; First posted 2015-06-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): People without keratoconus, history of ocular surgery, and other diseases mentioned in exclusion criteria. Normal people will receive treatment or measurement including: Schiotz tonometer measurement, UVA/riboflavin corneal crosslinking, Keratoplasty, Ocular morphology measurement,and routine ophthalmic examination.
  Interventions: Device: Schiotz tonometer; Device: UVA/riboflavin; Device: femto-LASIK; Device: Tomey SP-100 Pchymeter , Topolyzer Vario; Device: Topcon CT-80, Topcon, Japan; Device: Corvis-ST
- Keratoconic patients (Experimental): Patients with keratoconus.Keratoconic patients will receive treatment or measurement including:Schiotz tonometer measurement, UVA/riboflavin corneal crosslinking,Ocular morphology measurement,and routine ophthalmic examination.
  Interventions: Device: Schiotz tonometer; Device: UVA/riboflavin; Device: Tomey SP-100 Pchymeter , Topolyzer Vario; Device: Topcon CT-80, Topcon, Japan; Device: Corvis-ST
- Patients received keratoplasty (Experimental): Patients received keratoplasty. Patients received keratoplasty will receive treatment or measurement including:Schiotz tonometer measurement,Keratoplasty, Ocular morphology measurement,and routine ophthalmic examination..
  Interventions: Device: Schiotz tonometer; Device: femto-LASIK; Device: Tomey SP-100 Pchymeter , Topolyzer Vario; Device: Topcon CT-80, Topcon, Japan; Device: Corvis-ST

INTERVENTIONS:
Device: Schiotz tonometer — The corneal biomechanical properties will be measured using a Schiotz tonometer with routine manipulation protocol.This measurement will be used in normal people, keratoconic patients, patients received keratoplasty.
Device: UVA/riboflavin — The UVA/riboflavin corneal crosslinking will be applied using a UV-X lamp (Peschke Meditrade GmbH, Switzerland) with routine manipulation protocol (3mW/cm2, 365nm, 30 minutes).This treatment will be used in keratoconic patients.
  Arms: Control; Keratoconic patients
Device: femto-LASIK — The keratoplasty mainly include femto-LASIK (Laser in situ keratomileusis), which will be applied using a Wavelight FS200 and Wavelight EX500 Excimer Laser (Alcon Inc. USA.).The keratoplasty will be applied in patients who would like to receive the surgery.
  Arms: Control; Patients received keratoplasty
Device: Tomey SP-100 Pchymeter , Topolyzer Vario — Cornea thickness will be measured with a pachymeter (Tomey SP-100 Pchymeter, Japan); cornea topography will be measured with Topolyzer Vario (Allegro, Wavelight GmBH, Germany); anterior chamber depth, white to white, and ocular axis length will be measured using a IOL master (Carl Zeiss Meditec, Germany). These measurements will be used in normal people, keratoconic patients, patients received keratoplasty.
Device: Topcon CT-80, Topcon, Japan — Vision acuity will be measured with a decimal visual chart; IOP (Intra-ocular pressure) will be measured with a tonometer (Topcon CT-80, Topcon, Japan) , fundoscopy examination will be apllied with a direct ophthalmoscopy, slit lamp examination will be applied with a slit lamp. These examinations will be used in normal people, keratoconic patients, patients received keratoplasty.
Device: Corvis-ST — Cornea biomechanical properties will be measured with a ocular response analyzer (Reichert, USA.) and/or a Corvis-ST (Oculus, Germany).These measurements will be used in normal people, keratoconic patients, patients received keratoplasty.

SUMMARY:
This study aims to use Schiotz tonometer to evaluate the corneal biomechanical properties. The administration of Schiotz tonometer is according to the routine protocol which is use to measure intra-ocular pressure. The results obtained from Schiotz tonometer will be compared with results obtained from ORA and/or Corvis.

DETAILED DESCRIPTION:
Schiotz tonometer, since it firstly be developed more than 100 years ago by Hjalmar Schiotz, has been regarded as a classical method to evaluate intraocular pressure (IOP). In present study, we aims to measure the corneal biomechanical properties with schiotz tonometer and elucidate the clinical significance of this novel measurement. The corneal biomechanical property was calculated with subtracting the value displayed under loaded weight 5.5g from that under loaded weight 7.5g. We named the corneal biomechanical properties obtained with schiotz tonometer as Mulee factor, and the formulation is Mulee factor=value under loaded weight 7.5g (Value 7.5G)-value under loaded weight 5.5g (Value 5.5G).

ELIGIBILITY:
Inclusion Criteria:

* People without the disease mentioned in exclusion criteria part.

Exclusion Criteria:

* Patients with ocular diseases including keratitis, conjunctivitis, history of chronic eye/systemic diseases except myopia and keratoconus, history of ocular surgery except LASIK, pregnant or lactating females.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The Mulee factor obtained with Schiotz tonometer as a measure of cornea biomechanical property | up to 1 year
  Mulee factor= Value displayed with Schiotz tonometer under 7.5g load-Value displayed with Schiotz tonometer under 5.5g load

CONTACTS AND LOCATIONS:
Overall Officials: Guoying Mu, MD., Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China